CLINICAL TRIAL: NCT01752985
Title: A Double-Blind, Placebo-Controlled, Randomized, Two-stage, Parallel-Group, Adaptive Design Phase 2a Study to Evaluate the Effects of BMS-813160 in Subjects With Type 2 Diabetes Mellitus and Diabetic Kidney Disease (DKD) Who Have Residual Macroalbuminuria Despite Treatment With an Inhibitor of the Renin-Angiotensin System
Brief Title: Study to Evaluate the Effects of BMS-813160 on Protein Loss in the Urine of Subjects With Type 2 Diabetes and Diabetic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV202-010; 2012-005093-54 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2012-12-19 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — BMS-813160

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A: BMS-813160 150 mg & Placebo matching with BMS-813160 (Experimental): BMS-813160 150 mg capsules by mouth in AM and Placebo matching with BMS-813160 in PM for 12 weeks
  Interventions: Drug: BMS-813160; Drug: Placebo matching with BMS-813160
- Arm B: BMS-813160 300 mg (Experimental): BMS-813160 300 mg capsules by mouth twice daily for 12 weeks
  Interventions: Drug: BMS-813160
- Arm C: Placebo matching with BMS-813160 (Placebo Comparator): Placebo matching with BMS-813160 0 mg capsules by mouth twice daily for 12 weeks
  Interventions: Drug: Placebo matching with BMS-813160

INTERVENTIONS:
Drug: BMS-813160
  Arms: Arm A: BMS-813160 150 mg & Placebo matching with BMS-813160; Arm B: BMS-813160 300 mg
Drug: Placebo matching with BMS-813160
  Arms: Arm A: BMS-813160 150 mg & Placebo matching with BMS-813160; Arm C: Placebo matching with BMS-813160

SUMMARY:
The purpose of this study is to determine whether BMS-813160 will reduce the amount of protein loss in the urine of subjects with type 2 diabetes and diabetic kidney disease

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes mellitus with macroalbuminuria (UACR between 200 and 3500 mg/g)
* Background angiotensin converting enzyme inhibitor (ACEI) or angiotensin-receptor blocker (ARB) therapy

Exclusion Criteria:

* Clinical diagnosis of type 1 diabetes
* Unstable cardiovascular, metabolic, or other chronic disease status
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2
* High risk of infection or immune compromise
* Clinically significant ECG conduction abnormalities
* Drugs with significant potential to affect BMS-813160 exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (41):
  - Uab Hospital, Birmingham, Alabama
  - Univ Of Al At Birmingham, Birmingham, Alabama
  - Akdhc Medical Research Services Llc, Phoenix, Arizona
  - Academic Medical Research Institute, Los Angeles, California
  - Ucla, Los Angeles, California
  - Providence Clinical Research, North Hollywood, California
  - Diabetes Medical Center Of California, Northridge, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - All Medical Research, Llc, Cooper City, Florida
  - International Research Associates, Llc, Hialeah, Florida
  - Genesis Clinical Research, Inc., Tampa, Florida
  - Emory University School Of Medicine, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - John H. Stroger, Jr. Hospital Of Cook County, Chicago, Illinois
  - Research By Design, Llc, Evergreen Park, Illinois
  - St Louis Center Clinl Res, St Louis, Missouri
  - St. Louis Center For Clinical Research, St Louis, Missouri
  - Va Nebraska-Western Iowa Health Care System (Nwihcs), Omaha, Nebraska
  - Southern Nh Diab And Endo, Nashua, New Hampshire
  - Premier Research, Inc., Trenton, New Jersey
  - Albany Medical College, Albany, New York
  - The Endocrine Group Llp, Albany, New York
  - Nephrology Associates, Flushing, New York
  - Medispect Medical Research, Llc, Boone, North Carolina
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Piedmont Health Grp, Llc-Twr Pt Res Ctr, Hodges, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Doctors Hospital At Renaissance, Edinburg, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Northeast Clinical Research Of San Antonio, Llc, Schertz, Texas
  - Burke Internal Medicine And Research, Burke, Virginia
  - Virginia Endocrinology Research, Chesapeake, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Mcguire Va Medical Center, Richmond, Virginia
- Canada (9):
  - Health Sciences Centre Diabetes Research Centre, Winnipeg, Manitoba
  - Eastern Health Sciences Center, St. John's, Newfoundland and Labrador
  - Aggarwal And Associates, Brampton, Ontario
  - Clinical Research Solutions, Inc, Kitchener, Ontario
  - Lmc Diabetes & Endocrinology (Thornhill), Thornhill, Ontario
  - Lmc Diabetes & Endocrinology (Bayview), Toronto, Ontario
  - Centre De Recherche Clinique De Laval, Laval, Quebec
  - Recherche Gcp Research, Montreal, Quebec
  - Local Institution, Montreal, Quebec
- Denmark (4):
  - Local Institution, Frederiksberg
  - Local Institution, Gentofte Municipality
  - Local Institution, Hillerød
  - Local Institution, Holstebro
- France (6):
  - Local Institution, Amiens
  - Local Institution, Grenoble
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Tours

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 319 were enrolled, 110 completed screening, rest 209 discontinued: (Main reason:did not meet study criteria). Of 110 screened, 98 entered Placebo Lead-in period of which 89 completed period, rest 9 discontinued (2 due to Admin. reason, 3 no longer met study criteria, 2 AEs and 2 were lost to follow-up.)1 was randomized but declined treatment
Groups:
- BMS-813160 150 mg QD: Participants received BMS-813160 150 mg, capsule, orally along with matching placebo in Ante Meridiem (AM) and 2 Placebo matching with BMS-813160, capsules, orally in Post Meridiem (PM) for 12 weeks. Participants were followed up for 4 weeks post treatment.
- BMS-813160 300 mg BID: Participants received 2 BMS-813160 150 mg capsules, orally, twice daily (2*150 in AM and 2*150 in PM) for 12 weeks. Participants were followed up for 4 weeks post treatment.
- Placebo: Participants received BMS-813160 matching placebo capsules, orally, twice daily in AM and PM for 12 weeks and were followed up for 4 weeks post treatment.
Period: Treatment Period
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Started | 29 | 30 | 29
Completed | 25 | 27 | 24
Not Completed | 4 | 3 | 5
Not completed — Subject request to discontinue treatment | 1 | 0 | 1
Not completed — Subject no longer meets study criteria | 0 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Follow-up Period
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Started | 28 (Includes 25 participants in this period and 3 participants re-joined for follow-up) | 27 | 26 (Includes 24 participants in this period and 2 participants re-joined for follow-up)
Completed | 28 | 27 | 26
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 29 | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (9.58) | 60.2 (8.31) | 60.6 (11.52) | 61.5 (9.90)
Age, Customized [Number; unit: Participants]
  <65 years | 14 | 17 | 17 | 48
  >=65 years | 15 | 13 | 12 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 8 | 17
  Male | 27 | 23 | 21 | 71

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Urinary Albumin-to-Creatinine Ratio (UACR) Across 12 Weeks of Treatment With BMS-813160
Description: The presence of albumin in the urine (macroalbuminuria) is a marker of kidney disease. Albumin and creatinine concentrations were obtained from spot urine samples. UACR was calculated as the geometric mean of two first-morning void urine UACR measurements with samples collected on two separate occasions within a 4-day period.
Time Frame: Baseline, Weeks 2, 4, 8, 12, and 16 (Follow-up)
Population: The analysis was performed in all the participants who received any study drug. Here, 'n' signifies evaluable participants for specified categories in respective treatment arms.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 29 | 30 | 29
Percent Change
  Week 2: number analyzed (Participants) | 28 | 27 | 28
  Week 2 | 5.78 (48.994) | 3.79 (62.795) | 2.05 (30.771)
  Week 4: number analyzed (Participants) | 28 | 26 | 28
  Week 4 | 18.43 (62.661) | 5.81 (83.274) | 1.46 (40.051)
  Week 8: number analyzed (Participants) | 26 | 26 | 26
  Week 8 | 19.49 (65.381) | 9.87 (56.557) | 5.68 (43.659)
  Week 12: number analyzed (Participants) | 22 | 26 | 24
  Week 12 | 6.91 (56.666) | 29.16 (78.69) | 8.91 (54.025)
  Week 16: number analyzed (Participants) | 26 | 30 | 23
  Week 16 | 0.97 (61.72) | 20.63 (85.578) | 23.77 (70.411)

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Who Died and With Other (Not Including Serious) Adverse Events
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, or a congenital anomaly, or a medically important event.
Time Frame: From the date of subject's written consent until 30 days post discontinuation of dosing, assessed up to 26 months
Population: The analysis was performed in all the participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 29 | 30 | 29
Participants
  SAEs | 3 | 3 | 1
  Death | 0 | 1 | 0
  Other (Non-Serious) Adverse Events 5 % cut-off | 3 | 2 | 4

3. Secondary Outcome: Number of Participants With Out-of-Range Electrocardiogram (ECG) Interval
Description: 12-lead ECGs were performed before and 1 hour after dosing at Weeks 0, 2 and 4. ECGs were recorded after the participant has been supine for at least 5 minutes. The PR interval was defined as the beginning of the P wave to the beginning of the QRS complex, and represents the time taken by electrical impulse to travel from the sinus node through the atrioventricular (AV) node. The QRS complex represented the rapid depolarization of the right and left ventricles. The QT interval was defined as the time from the start of the Q wave to the end of the T wave, and represents the time taken for ventricular depolarization and repolarization. Participants were evaluated for abnormal ECG intervals. Criteria's for abnormality were PR >200, QRS >120, QT >500, QTcF >450, Change From Baseline >30 milliseconds (msec).
Time Frame: Baseline up to Week 16
Population: The analysis was performed in all the participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 29 | 30 | 29
Participants
  PR >200 msec | 8 | 8 | 4
  QRS >120 msec | 3 | 3 | 3
  QT >500 msec | 0 | 1 | 0
  QTcF >450 msec | 7 | 5 | 6
  Change from baseline in QT >30 msec | 8 | 6 | 4
  Change from baseline in QTcF >30 msec | 4 | 3 | 1

4. Secondary Outcome: Trough Observed Plasma Concentration (Ctrough) of BMS-813160
Description: Ctrough is the minimum estimated plasma concentration at steady state.
Time Frame: Pre-dose at Week 2, 4, 8, 12 and 0.5, 1, 2, 4, and 6 hours post-dose at Week 12
Population: The analysis was planned to be performed in the Pharmacokinetic (PK) analysis set which included all participants who receive a dose of study drug and have adequate PK concentration-time data. Data was not collected for any participants due to termination of the study
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Area Under The Plasma Concentration-Time Curve From Time Zero to 6 Hours Post-Dose [AUC(0-6 h)]
Description: AUC(0-6 h) is the area under the plasma concentration-time curve from pre-dose (0 h) to 6 h post-dose.
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Week 12
Population: as for outcome 4
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Renal Clearance (CLr) of BMS-813160
Description: CLr was calculated by dividing the total amount excreted in the urine from 0 to 6 hours by the area under the plasma concentration-time curve from time zero extrapolated to infinite time. The renal function was classified based on estimated glomerular filtration rate as normal (>=90 mL/min/1.73 m^2), mildly impaired (60-89 mL/min/1.73 m^2), moderately impaired stage 3A (45-59 mL/min/1.73 m^2), and moderately impaired stage 3B (30-44 L/min/1.73 m^2).
Time Frame: Pre-dose, 0.5, 1, 2, 4, and 6 hours post-dose at Week 12
Population: The analysis was planned to be performed in the Pharmacokinetic (PK) analysis set which included all participants who receive a dose of study drug and have adequate PK concentration-time data.Data was not collected for any participants due to termination of the study
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Dose-Response Relationship Using Change in Baseline Urinary Albumin-to-Creatinine Ratio (UACR) Across 12 Weeks of Treatment
Description: The presence of albumin in the urine (macroalbuminuria) is a marker of kidney disease. Albumin and creatinine concentrations were obtained from spot urine samples. UACR was calculated as the geometric mean of two first-morning void urine UACR measurements with samples collected on two separate occasions within a 4-day period. The effect of BMS-813160 on urinary albumin excretion as measured by UACR values in participants with diabetic kidney disease after 12 weeks of treatment was assessed. The model included treatment group as a main effect, and the log of baseline UACR values, as well as baseline values of eGFR, blood pressure, blood glucose and lipid levels, as covariates.
Time Frame: Baseline, Weeks 2, 4, 8 and 12
Population: Data was not collected for any participants due to termination of the study
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of participant's written consent until 30 days post discontinuation of dosing, assessed up to 26 months
Groups:
- BMS-813160 300 mg BID: Participants received 2 BMS-813160 150 mg capsules, orally, twice daily (2*150 in AM and 2*150 in PM) for 12 weeks.
- Placebo: Participants received BMS-813160 matching placebo capsules, orally, twice daily in AM and PM for 12 weeks.
Arm/Group | BMS-813160 150 mg QD | BMS-813160 300 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 1/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 3/29 | 3/30 | 1/29
Other Adverse Events (participants affected / at risk) | 3/29 | 2/30 | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-813160 150 mg QD (N=29) | BMS-813160 300 mg BID (N=30) | Placebo (N=29)
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-813160 150 mg QD (N=29) | BMS-813160 300 mg BID (N=30) | Placebo (N=29)
Oedema peripheral (General disorders) | 1 | 2 | 3
Fatigue (General disorders) | 3 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.